CLINICAL TRIAL: NCT05852912
Title: Effects on Physical and Mental Prognosis and Quality of Life of Elderly People With Depressive Symptoms: Development of Wearable Devices and Telemedicine as Assessment Tools
Brief Title: Effects on Physical and Mental Prognosis and Quality of Life of Elderly People With Depressive Symptoms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200501B0C603
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Depression
Keywords: Elderly; wearable devices
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- elders combined with mild mental illness: elders combined with mild mental illness(120 subjects)
- elders combined without mild mental illness: elders combined without mild mental illness(120 subjects)

SUMMARY:
Mild mental illnesses such as depression, anxiety, and sleep disorders in the elderly are also major health issues for Taiwanese. Mild mental illnesses that cannot be effectively treated may worsen existing chronic diseases. However, there is a lack of objective, convenient and effective assessment tools for the cognitive, emotional, sleep and other mental health of the elderly. The development of these assessment tools can be used to quantify the degree of abnormality, provide early diagnosis, and evaluate the effectiveness of long-term care.

In recent years, the progress of physiological sensing technology and wearable devices,telemedicine devices and various computer information integration software has provided objective clinical data. This study will use "wearable devices", "telemedicine" and "computer information software" to evaluate whether elderly with mild mental illness have a poor prognosis. In this way, an intelligent care model for "cognitive, emotional, sleep and other mental health" for elderly is developed.

DETAILED DESCRIPTION:
Mild mental illnesses such as depression, anxiety, and sleep disorders in the elderly are also major health issues for Taiwanese. Mild mental illnesses that cannot be effectively treated may worsen existing chronic diseases. However, there is a lack of objective, convenient and effective assessment tools for the cognitive, emotional, sleep and other mental health of the elderly. The development of these assessment tools can be used to quantify the degree of abnormality, provide early diagnosis, and evaluate the effectiveness of long-term care.

In recent years, the progress of physiological sensing technology and wearable devices,telemedicine devices and various computer information integration software has provided objective clinical data. This study will use "wearable devices", "telemedicine" and "computer information software" to evaluate whether elderly with mild mental illness have a poor prognosis. In this way, an intelligent care model for "cognitive, emotional, sleep and other mental health" for elderly is developed.

This study is expected to have the following objectives:

1. To understand the prevalence and current situation of Taiwanese elderly complicated with mild mental illnesses (such as anxiety, insomnia, etc.).
2. Establish a physical and mental assessment tool for the elderly, integrating different scales such as physical health, mental health, and mobility into a complete and convenient information interface for the elderly, caregivers, and medical staff to use to facilitate cross-field connections Communities and hospitals, providing continuum of care.
3. Introduce wearable devices and computerized software to analyze the prognosis of elderly hypertensive patients.

Through this project, it is expected to combine the two majors of medical treatment and information technology, and integrate various assessment tools into a convenient information interface, making it easy for the elderly and caregivers to use, and even linking to the medical network to assist in rapid diagnosis, referral and receive treatment. The collected data can be used for big data analysis in the future to provide further national policy reference.

ELIGIBILITY:
Inclusion Criteria:

1. Age is more than or equal to 65 years old
2. Able to provide informed consent to participate in the research.
3. Can understand the instructions, and coduct the questionnaire assessment and physical function measurement.

Exclusion Criteria:

1. Those unable to give consent to participate in the research.
2. Those who cannot understand the instructions, difficult to coduct questionnaire assessment and physical function measurement.
3. Severe disease state (respiratory distress requiring intubation or patient with terminal illness) or severe brain injury or severe Dementia.
4. Snstable patients and patients with substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The elderly who's age is more than or equal to 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Actigraphy | Four times a year until the study is completed (up to 3 years)
  Change in sleep latency (mins) based on actigraphy during the study.

SECONDARY OUTCOMES:
Actigraphy-SOL | Four times a year until the study is completed (up to 3 years)
  sleep onset latency (SOL)based on actigraphy during the study.
Actigraphy-TST | Four times a year until the study is completed (up to 3 years)
  Total sleep time (TST, mins) based on actigraphy during the study.
Actigraphy-SE | Four times a year until the study is completed (up to 3 years)
  Sleep efficiency (SE, %) based on actigraphy during the study.
Actigraphy-WASO | Four times a year until the study is completed (up to 3 years)
  Wake after sleep onset (WASO) based on actigraphy during the study.
Actigraphy-Awake time | Four times a year until the study is completed (up to 3 years)
  Awake time based on actigraphy during the study.
Actigraphy-TIB | Four times a year until the study is completed (up to 3 years)
  Time in bed(TIB) based on actigraphy during the study.
Conners' Continuous Performance Test (CPT) | Four times a year until the study is completed (up to 3 years)
  The Conners Continuous Performance Test is a computer administered test that is designed to assess problems with attention,impulsivity and vigilance .Many statistics are computed including omission errors , commission errors, hit reaction time, hit reaction time standard error, detectability, response style, perseverations , hit reaction time by block, standard error by block, reaction time by ISI , and standard error by ISI. These statistics are converted to T-scores and can be interpreted in terms of various aspects of attention including inattention, impulsivity, and vigilance.Higher rates of correct detections indicate better attentional capacity.
Epworth Sleepoiness Scale (ESS) | Four times a year until the study is completed (up to 3 years)
  Epworth Sleepoiness Scale (ESS) assesses the responder's propensity to doze or fall asleep during 8 common daily activities, such as: sitting and reading; sitting inactive in a public place; sitting and talking to someone; sitting quietly after a lunch without alcohol; or in a car, while stopped for a few minutes in traffic.
  Score of 0 to 10 indicate normal range of sleepiness in healthy adults.;11 to 14 indicate mild sleepiness;15 to 17 indicate moderate sleepiness;18 to 24 indicate severe sleepiness .
Short Form-36 (SF-36) | Four times a year until the study is completed (up to 3 years)
  36-Item Short-Form Health Survey (SF-36) includes 11 major questions that evaluate eight components (0-100), with higher scores indicating better outcome.These components include physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional wellbeing, social functioning, pain, and general health.
Geriatric Depression Scale-15(GDS-15) | Four times a year until the study is completed (up to 3 years)
  The Geriatric Depression Scale-15 is a screening tool used to identify symptoms of depression in elderly adults.Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.It takes about 5 to 7 minutes to complete.
Montreal Cognitive Assessment (MoCA) | Four times a year until the study is completed (up to 3 years)
  The Montreal Cognitive Assessment is a test used by healthcare providers to evaluate people with memory loss or other symptoms of cognitive decline. It can help identify those at risk for developing Alzheimer's disease and other forms of dementia. It is also used as a screening tool for conditions like Parkinson's disease, brain tumors, substance abuse, and head trauma.
  The MoCA checks different types of cognitive or thinking abilities. These include:orientation,short-term memory/delayed recall,executive function/visuospatial ability,language,abstraction,naming,attention.
  Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.1 point is added to the test-taker's score if they have 12 years or less of formal education.
  The MoCA contains 30 questions and takes around 10 to 12 minutes to complete.
Hospital Anxiety and Depression Scale(HADS) | Four times a year until the study is completed (up to 3 years)
  The Hospital Anxiety and Depression Scale aims to measure symptoms of anxiety and depression.As in the HADS, the response to each item is rated 0-3. Higher scores indicate higher levels of anxiety or depression.
Pittsburgh Sleep Quality Index (PSQI) | Four times a year until the study is completed (up to 3 years)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire for assessing the subjective sleep quality, which consists of 19 items and can be calculated and combined into 7 clinically-derived component score (0-3), with higher scores indicating worse sleep quality.
Activities of Daily Living (ADL) | Four times a year until the study is completed (up to 3 years)
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.Scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-100 indicates "slight" dependency.
Lawton Instrumental Activities of Daily Living Scale (IADL) | Four times a year until the study is completed (up to 3 years)
  The Instrumental Activities of Daily Living (IADL) Scale is used to assess independent living skills of an individual and measures functional ability as well as declines and improvements over time. The test measures eight realms of function through self report, which attempt to assess everyday functional competence in the elderly. This is done by evaluating a more complex set of behaviours like telephoning, shopping, food preparation, housekeeping, laundering, use of transportation, use of medicine, and financial behaviour. Each domain measured by the scale relies on either cognitive or physical function, though all require some degree of both.
  The Lawton IADL scale can be scored in several ways, the most common method is to rate each item either dichotomously (0 = less able, 1 = more able) or trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the eight responses. The higher the score, the greater the person's abilities.
Insomnia Severity Index(ISI) | Four times a year until the study is completed (up to 3 years)
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia.The usual recall period is the "last month" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Clinical Frailty Scale (CFS) | Four times a year until the study is completed (up to 3 years)
  The clinical frailty scale is a 9-point scale that quantifies frailty based on function in individual patients. It is complemented by a visual chart to assist with the classification of frailty. Higher scores indicate increased frailty and associated risks.

OTHER OUTCOMES:
Heart rate variability (HRV) device | Four times a year until the study is completed (up to 3 years)
  The measurement method is to stick four patches on participants body and measure the heart rhythm state for 10 minutes. An estimate was computed for LF/HF ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shu Huang, Study Director — Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blood ML, Sack RL, Percy DC, Pen JC. A comparison of sleep detection by wrist actigraphy, behavioral response, and polysomnography. Sleep. 1997 Jun;20(6):388-95. PMID 9302721
- [Result] Chen NH, Johns MW, Li HY, Chu CC, Liang SC, Shu YH, Chuang ML, Wang PC. Validation of a Chinese version of the Epworth sleepiness scale. Qual Life Res. 2002 Dec;11(8):817-21. doi: 10.1023/a:1020818417949. PMID 12482165
- [Result] Chu KC, Huang YS, Tseng CF, Huang HJ, Wang CH, Tai HY. Reliability and validity of DS-ADHD: A decision support system on attention deficit hyperactivity disorders. Comput Methods Programs Biomed. 2017 Mar;140:241-248. doi: 10.1016/j.cmpb.2016.12.003. Epub 2016 Dec 16. PMID 28254080
- [Result] Edd EM, Flores S. Sleepiness or excessive daytime somnolence. Geriatr Nurs. 2009 Jan-Feb;30(1):53-60. doi: 10.1016/j.gerinurse.2008.11.004. PMID 19215814
- [Result] Hegerl U, Wilk K, Olbrich S, Schoenknecht P, Sander C. Hyperstable regulation of vigilance in patients with major depressive disorder. World J Biol Psychiatry. 2012 Sep;13(6):436-46. doi: 10.3109/15622975.2011.579164. Epub 2011 Jul 4. PMID 21722018
- [Result] Huang YL, Liu RY, Wang QS, Van Someren EJ, Xu H, Zhou JN. Age-associated difference in circadian sleep-wake and rest-activity rhythms. Physiol Behav. 2002 Aug;76(4-5):597-603. doi: 10.1016/s0031-9384(02)00733-3. PMID 12126998
- [Result] Hung CI, Weng LJ, Su YJ, Liu CY. Depression and somatic symptoms scale: a new scale with both depression and somatic symptoms emphasized. Psychiatry Clin Neurosci. 2006 Dec;60(6):700-8. doi: 10.1111/j.1440-1819.2006.01585.x. PMID 17109704
- [Result] Ismail Z, Gatchel J, Bateman DR, Barcelos-Ferreira R, Cantillon M, Jaeger J, Donovan NJ, Mortby ME. Affective and emotional dysregulation as pre-dementia risk markers: exploring the mild behavioral impairment symptoms of depression, anxiety, irritability, and euphoria - CORRIGENDUM. Int Psychogeriatr. 2019 Jan;31(1):157. doi: 10.1017/S1041610218000637. Epub 2018 Nov 21. No abstract available. PMID 30461372
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Kemp AH, Quintana DS, Felmingham KL, Matthews S, Jelinek HF. Depression, comorbid anxiety disorders, and heart rate variability in physically healthy, unmedicated patients: implications for cardiovascular risk. PLoS One. 2012;7(2):e30777. doi: 10.1371/journal.pone.0030777. Epub 2012 Feb 15. PMID 22355326
- [Result] Kok RM, Reynolds CF 3rd. Management of Depression in Older Adults: A Review. JAMA. 2017 May 23;317(20):2114-2122. doi: 10.1001/jama.2017.5706. PMID 28535241
- [Result] Kim J, Nakamura T, Kikuchi H, Sasaki T, Yamamoto Y. Co-variation of depressive mood and locomotor dynamics evaluated by ecological momentary assessment in healthy humans. PLoS One. 2013 Sep 13;8(9):e74979. doi: 10.1371/journal.pone.0074979. eCollection 2013. PMID 24058642
- [Result] Lin C, Chin WC, Huang YS, Chu KC, Paiva T, Chen CC, Guilleminault C. Different circadian rest-active rhythms in Kleine-Levin syndrome: a prospective and case-control study. Sleep. 2021 Sep 13;44(9):zsab096. doi: 10.1093/sleep/zsab096. PMID 33851710
- [Result] Musiek ES, Bhimasani M, Zangrilli MA, Morris JC, Holtzman DM, Ju YS. Circadian Rest-Activity Pattern Changes in Aging and Preclinical Alzheimer Disease. JAMA Neurol. 2018 May 1;75(5):582-590. doi: 10.1001/jamaneurol.2017.4719. PMID 29379963
- [Result] Olbrich S, Sander C, Minkwitz J, Chittka T, Mergl R, Hegerl U, Himmerich H. EEG vigilance regulation patterns and their discriminative power to separate patients with major depression from healthy controls. Neuropsychobiology. 2012 Jun;65(4):188-94. doi: 10.1159/000337000. Epub 2012 Apr 26. PMID 22538271
- [Result] Olbrich S, van Dinteren R, Arns M. Personalized Medicine: Review and Perspectives of Promising Baseline EEG Biomarkers in Major Depressive Disorder and Attention Deficit Hyperactivity Disorder. Neuropsychobiology. 2015;72(3-4):229-40. doi: 10.1159/000437435. Epub 2016 Feb 23. PMID 26901357
- [Result] Ong AD, Uchino BN, Wethington E. Loneliness and Health in Older Adults: A Mini-Review and Synthesis. Gerontology. 2016;62(4):443-9. doi: 10.1159/000441651. Epub 2015 Nov 6. PMID 26539997
- [Result] Pan W, Song Y, Kwak S, Yoshida S, Yamamoto Y. Quantitative evaluation of the use of actigraphy for neurological and psychiatric disorders. Behav Neurol. 2014;2014:897282. doi: 10.1155/2014/897282. Epub 2014 Aug 19. PMID 25214709
- [Result] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Result] Sgoifo A, Carnevali L, Alfonso Mde L, Amore M. Autonomic dysfunction and heart rate variability in depression. Stress. 2015;18(3):343-52. doi: 10.3109/10253890.2015.1045868. Epub 2015 May 25. PMID 26004818
- [Result] Shaked D, Faulkner LMD, Tolle K, Wendell CR, Waldstein SR, Spencer RJ. Reliability and validity of the Conners' Continuous Performance Test. Appl Neuropsychol Adult. 2020 Sep-Oct;27(5):478-487. doi: 10.1080/23279095.2019.1570199. Epub 2019 Feb 22. PMID 30793982
- [Result] Stapelberg NJ, Hamilton-Craig I, Neumann DL, Shum DH, McConnell H. Mind and heart: heart rate variability in major depressive disorder and coronary heart disease - a review and recommendations. Aust N Z J Psychiatry. 2012 Oct;46(10):946-57. doi: 10.1177/0004867412444624. Epub 2012 Apr 23. PMID 22528974
- [Result] van Someren EJ, Hagebeuk EE, Lijzenga C, Scheltens P, de Rooij SE, Jonker C, Pot AM, Mirmiran M, Swaab DF. Circadian rest-activity rhythm disturbances in Alzheimer's disease. Biol Psychiatry. 1996 Aug 15;40(4):259-70. doi: 10.1016/0006-3223(95)00370-3. PMID 8871772
- [Result] Wahl D, Solon-Biet SM, Cogger VC, Fontana L, Simpson SJ, Le Couteur DG, Ribeiro RV. Aging, lifestyle and dementia. Neurobiol Dis. 2019 Oct;130:104481. doi: 10.1016/j.nbd.2019.104481. Epub 2019 May 25. PMID 31136814
- [Result] Wong NM, Liu HL, Lin C, Huang CM, Wai YY, Lee SH, Lee TM. Loneliness in late-life depression: structural and functional connectivity during affective processing. Psychol Med. 2016 Sep;46(12):2485-99. doi: 10.1017/S0033291716001033. Epub 2016 Jun 22. PMID 27328861
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820